CLINICAL TRIAL: NCT01665820
Title: Study EM-05-012530 Benefit of Auscultation With 3M™ Littmann® 3200 Electronic Stethoscope to Diagnose Murmurs and Heart Pathologies in Overweight and Obese Patients With Increased Layers of Adipose Tissue
Brief Title: Auscultate Obese Patients Using Electronic and Traditional Stethoscopes
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: Study EM-05-012530
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Chest Pathology
Keywords: chest; pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Auscultate with mechanical stethoscope: Cardiologist & Medical Resident auscultate using mechanical stethoscope
  Interventions: Device: Auscultate with electronic or mechanical stethoscope (3M Littmann)
- Auscultate with electronic stethoscope: Cardiologist & Medical Resident auscultate using electronic stethoscope
  Interventions: Device: Auscultate with electronic or mechanical stethoscope (3M Littmann)

INTERVENTIONS:
Device: Auscultate with electronic or mechanical stethoscope (3M Littmann)
  Other Names: 3M Littmann 3200 Electronic Stethoscope; 3M Littman Cardiology III Mechanical Stethoscope

SUMMARY:
Auscultating Obese patients using the 3M Littmann Electronic Model 3200 Stethoscope is more effective in identifying referrable murmurs than using a traditional stethoscope.

DETAILED DESCRIPTION:
Study will enroll subjects who have greater than 30 BMI ratings. Each subject will receive 4 auscultation examinations. Two auscultations will be done by a cardiologist using both an acoustic traditional stethoscope and an electronic stethoscope. Two additional auscultations will be done by a 3rd year medical resident also using both an acoustic traditional stethoscope and an electronic stethoscope. All determinations will be compared to echocardiography results.

ELIGIBILITY:
Inclusion Criteria:

* Greater or equal than 18 years of age
* Referred for an echocardiogram
* obese, as defined as having a BMI greater than 30
* volunteers to participate in study
* agrees to provide copy of echocardiogram exam report

Exclusion Criteria:

-Investigator believes subject should not be included or is unsuitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients greater or equal to 18 years of age, with a BMI greater than 30 and who have been scheduled for an echocadiogram examination
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Most severe cardiac lesion identified by auscultation & echocardiography | 0-4 days

SECONDARY OUTCOMES:
Secondary cardiac lesion identified by auscultation & echocardiography | 0 - 4 days
Other heart sounds identified by auscultation & echocardiography | 0 - 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Egle Kalinauskiene, MD, Study Director — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania